CLINICAL TRIAL: NCT01953016
Title: NIH Participation to USIDNET Registry
Brief Title: Participation in a Research Registry for Immune Disorders
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130199; 13-HG-0199
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Primary Immunodeficiencies; APECED; CGD; Wiskott-Aldrich Syndrome; SCID
Keywords: Job Syndrome/HIES; GATA2; Primary Immunodeficiency; SCID; DOCK8; Natural History
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune; Wiskott-Aldrich Syndrome; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- immunodeficiency: Individuals of all ages, gender, and races with an immunodeficiency disorder from NIH studies, will be accepted for registration.

SUMMARY:
Background:

- People with primary immune deficiency diseases (PIDD) have weak immune systems. This makes it hard for their bodies to fight infection. The Immune Deficiency Foundation has a network to collect data about people with PIDD. It is called the United States Immunodeficiency Network. It will help doctors and scientists better understand these disorders. The goal is to get medical data for everyone with these disorders in the U.S. and Canada. Data will be stored in a registry. Researchers can use it to study if these disorders are increasing. They can also learn how the disorders are diagnosed and treated.

Objectives:

- To collect data on people with primary immune deficiency disorders.

Eligibility:

- People who have a PIDD.

Design:

* Data can be added with no record of personal identity.
* Data can be added with identity kept separate. This data will be linked to the registry by a code number.
* Data for the registry includes:
* Family history
* Disease treatment
* Disease characteristics
* Medical history
* Laboratory data

DETAILED DESCRIPTION:
The purpose of this protocol is to provide a resource for clinical and laboratory research through enrollment of known immunodeficiency patients into a national registry, the US Immunodeficiency Network (USIDNET). The registry data will expand NIH s and the nation s knowledge base about immune deficiency disorders and genetic mutations that lead to these disorders. Additional registrants from NIH protocols will not only increase the understanding of the molecular basis of these disorders, but also will serve to document and track the incidence and progression of complications.

Objectives and specific aims

The purpose of this proposal is to create a mechanism for depositing NIH data into USIDNET. The patient Registry is designed to obtain longitudinal data on a large number of patients with primary immunodeficiency diseases, and genetic carriers of these defects in order to:

* Learn more about the phenotypic variations seen in a large number of individual patients with the same rare molecular diagnosis.
* Determine the natural history of these genetic disorders of immunity and establish genotype-phenotype correlations.
* Learn effects of various treatment protocols used in these patients over time, including unexpected side effects that may be unique to a particular diagnostic group.
* To evaluate quality of life using standard tools and correlate these with genotype and treatment history.
* To promote collaborative research amongst interested investigators by identifying a larger pool of potential research subjects than would be available at their own institutions
* To identify patients with a specific diagnosis for potential participation in multi-institutional clinical trials designed for diagnosis or therapy or their specific disease.

ELIGIBILITY:
* INCLUSION CRITERIA

Individuals of all ages, gender, and races with an immunodeficiency disorder from NIH studies will be accepted for registration. No healthy volunteers will be enrolled.

EXCLUSION CRITERIA

Individuals with immunodeficiency associated with HIV infection, chemotherapy or other immunosuppressive therapies will not be accepted for registration unless there is clear evidence that these individuals also have a genetically determined immunodeficiency disease as well. Adult individuals who do not give informed consent will also be excluded.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of all ages, gender, and races with an immunodeficiency disorder from NIH studies, will be accepted for registration.@@@
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Prevalence | Ongoing
  The Registry will provide a minimum estimate of the prevalence of each disorder in the US, a comprehensive clinical picture of each disorder, and a resource for clinical and laboratory research.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Garabedian, R.N., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ruffner MA; USIDNET Body Weight Group; Sullivan KE. Complications Associated with Underweight Primary Immunodeficiency Patients: Prevalence and Associations Within the USIDNET Registry. J Clin Immunol. 2018 Apr;38(3):283-293. doi: 10.1007/s10875-018-0492-0. Epub 2018 Apr 4. PMID 29619656
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-HG-0199.html